CLINICAL TRIAL: NCT05288920
Title: Effect of Pulsed Mode Radiofrequency on Dorsal Root Ganglion on Tumor Necrotic Factor α Level in Lumbar Disc Related Radicular Pain
Brief Title: Effect of Pulsed Mode Radiofrequency as a Treatment of Lumbar Disc Related Radicular Pain on Tumor Necrotic Factor α Level
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mona Hussein, Associate professor of Neurology, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMBSUREC/06042021/Fathy-1
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: To compare the effect of transforaminal injection of Steroids alone versus Radiofrequency pulsed mode on dorsal root ganglion combined with transforaminal steroids injection on TNF-α level in lumbar disc related radicular pain
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiofrequency group (Active Comparator): Radiofrequency pulsed mode on dorsal root ganglion combined with transforaminal steroids injection
  Interventions: Procedure: Radiofrequency pulsed mode on dorsal root ganglion combined with transforaminal steroids injection
- Steroids group (Placebo Comparator): Transforaminal injection of Steroids alone
  Interventions: Drug: Transforaminal injection of Steroids alone

INTERVENTIONS:
Procedure: Radiofrequency pulsed mode on dorsal root ganglion combined with transforaminal steroids injection — Radiofrequency pulsed mode on dorsal root ganglion combined with transforaminal steroids injection
  Arms: Radiofrequency group
Drug: Transforaminal injection of Steroids alone — Transforaminal injection of Steroids alone
  Arms: Steroids group

SUMMARY:
Lumbar radiculopathy is a term that describes symptoms of pain, numbness, and/or weakness that radiate along the sciatic nerve from the lower back to the buttocks and leg (1). Lumbar radiculopathy is a relevant health problem that affects quality of life, resulting in high health costs and economic loss worldwide (2). The reported prevalence of sciatica varies widely from 1.2% and 43% in the general population (3).

Although initially believed to be a primary mechanical insult to the nerve root and dorsal root ganglion, lumbar radiculopathy is possibly caused by inflammatory changes in the nerve root (4). The role of cytokine-mediated neuroimmune interactions in the development and persistence of pain has been extensively studied (5,6,7).

Intraneural application of pro-inflammatory cytokines induces behavioral signs associated with pain (8). Anti-inflammatory cytokine treatment effectively reduces hyperalgesia (9). Inflammatory cytokine inhibitors provided long-lasting analgesia in an inflammatory neuropathic pain model. On the basis of these findings, we evaluated whether cytokine profiles differ between severe and mild human sciatica, as well as whether distinct cytokine profiles provide relevant information regarding lumbar radiculopathy pathogenesis. (10,11).

Tumor necrosis factor-alpha (TNF-α) is a pleiotropic cytokine that can stimulate inflammatory responses of synapses and myelin sheath, promote cellular apoptosis because of its cytotoxic effect, and induce nerve swelling and neuropathic pain (12).

TNF-α influences neural survival, exerting both neuroprotective and neurodegenerative actions (13). Following peripheral nerve injury, upregulation of TNF-α expression has been documented in several neuropathic pain models (14).

Pulsed radiofrequency (PRF) is a relatively new developed technique that is a variation of conventional radiofrequency treatment. PRF treatment does not allow temperatures above 42°C at the tip of the electrode. PRF provides advantage avoiding thermal tissue destruction and pain sequelae in management of pain. Recently, it has been recommended for treatment of chronic pain (15).

Electromagnetic field which is thought to be responsible for the clinical effect of pulsed RF spread from active tip of electrode to around the electrode. The most intense part of the electromagnetic field is pointed tip of the electrode (16). It is a minimally invasive technique that involves application of electric fields to nerves to inhibit nociceptive stimuli and prevent pain transmission. PRF can be considered when conventional treatments have intolerable side effects or do not sufficiently relieve pain (17).

Working mechanism of PRF which is recently more preferred technique to treat chronic pain due to not forming tissue damage and less painful procedure is not exactly known but it is considered to act neuromodulation (18).

The aim of this work is to compare the effect of transforaminal injection of Steroids alone versus Radiofrequency pulsed mode on dorsal root ganglion combined with transforaminal steroids injection on TNF-α level in lumbar disc related radicular pain

DETAILED DESCRIPTION:
This is a prospective randomized controlled trial that will be carried out on 80 patients diagnosed as having symptomatic lumbar disc prolapse.

The study will be planned by taking the local ethics committee approval and patients' written consent. Between 20-75 years of age, 40 patients will receive pulsed radiofrequency on dorsal root ganglion combined with transforaminal steroids injection procedure and 30 patients will receive transforaminal steroid injection. All patients are suffering more than 3 months long chronic pain syndrome.

Patients will be informed about the technique, at the level of cooperation that can provide this information to understand and work with patients who have the level of cooperation that can provide this information to understand and agree to participate in work will be included in the study. Patients included in the study will be given an appointment for the procedure and Written consent will be obtained from all participants .The patients will be recruited from the neurology and pain clinic of Beni-Suef University Hospital, in the period from March 2022 to September 2022.

Inclusion criteria:

Patients diagnosed as having symptomatic lumbar disc prolapse based on the following:

1. Clinical evidence of disc pulge in the form of disc related radicular pain of >3 months duration, not responding to conservative treatment and interfering with daily activities
2. Radiological demonstration of posterolateral lumbar disc pulge by MRI lumbosacral
3. Age range is between 30-80 years

Exclusion criteria:

The following patients will be excluded from the study:

1. Patients with spinal deformities
2. Patients with a previous history of spinal trauma
3. Patients with previous spinal surgery
4. Patients with radiological evidence of any inflammatory or neoplastic lesion affecting the spinal cord or vertebral column
5. Patients with severe lumbar disc herniation causing lower limb weakness or sphincteric troubles
6. Patient with pain rather than radicular neuropathic pain as Facet osteoarthritis, Sacroiliitis, Hip osteoarthritis, Discogenic, Pyriformis syndrome.
7. Patients with contraindications to interventions (coagulopathy, sepsis, or allergy to the used drugs)
8. Patients with contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body).
9. Pregnant
10. History of G6PD deficiency in patients who are candidates to receive ozone therapy.
11. Suspected spondylodiscitis.

METHODS:

All patients will be subjected to the following:

1) Clinical assessment:

1. Detailed history taking regarding: duration of pain, the presence of discogenic pain, radicular pain, responseto medical treatment, or previous interventional pain management
2. Neurological examination: motor and sensory examination
3. Assessment of the severity of the neurological symptoms before and 2 weeks,1 and 3 months, after the interventional procedure by a physician who will be blinded to the type of intervention.

   Modified Oswestry Back Disability Score (MODI): It consisted of low back pain disability index questionnaire about pain intensity, personal care, lifting, standing, walking, sitting, sleeping, social life, travelling and employment/homemaking. Thus, total 10 points; each had score range of 0-5. Hence, total score had range of 0-50. A high MODI score indicates a more severe functional disability related to the pain.

   Numeric Rating Scale (NRS-11): It is a scale for assessment of intensity of pain. It ranged from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain.
4. Assessment of patient's satisfaction about the intervention 3 months after the interventional procedure by a physician who will be blinded to the patient's condition and the type of intervention.

The Short Assessment of Patient Satisfaction (SAPS): It consists of seven items assessing the core domains of patient satisfaction which include treatment satisfaction, explanation of treatment results, clinician care, participation in medical decision making, respect by the clinician, time with the clinician, and satisfaction with hospital/clinic care. Responses scales are 5-point scales. SAPS scores can be interpreted as follows: 0 to 10 = very dissatisfied, 11 to 18 = dissatisfied, 19 to 26 = satisfied, 27 to 28 = very satisfied.

2) Laboratory assessment: Blood samples will be collected for all included patients in a fasting state, before and three months after the interventional pain management. They will be centrifuged (2000 U/min) at 4C, and stored at 80C. Serum TNFα will be measured with a high-sensitivity TNFα Quantikine immunoassay.

3) Radiological assessment: Magnetic Resonance imaging of the lumbosacral spine will be performed for all patients included in the study.

Magnetic Resonance imaging (MRI):

The following protocols will be used:

1. T1- weighted images (axial, sagittal).
2. T2- weighted images (axial, coronal).
3. Fluid attenuated inversion recovery (FLAIR) sequence. 4) Interventional pain management: Patients will be randomly assigned into one of two groups. In all cases taken to the operating room, routine monitoring was conducted. ECG, noninvasive blood pressure and peripheral arterial saturation (SpO2) was monitored. After the monitoring, patients will be taken the convenient position for the procedure. The C-arm fluoroscopy will be used for imaging during process.

(1) Transforaminal steroid injection group: The selected patients will receive transforaminal epidural injection of premixed steroids with local anesthetic in a total volume 2 ml (7 mg Betamethasone and 20 mg Lidocaine 2%) (2) radiofrequency on dorsal root ganglion combined with transforaminal steroids injection group: The needle puncture site determined by fluoroscopy. The Radiofrequency (RF) application was performed to all patients as detailed below: following subcutaneous local anesthesic infiltration, Cosman RFG1A Lesion Generator (Cosman Medical, Inc., Burlington, Massachusetts, USA) was used for RF thermo-ablation.

RF cannula (22 g, 10 cm, 5 mm active electrode tip or 5 cm, 2 mm active electrode tip) was placed in a determined puncture site before processing and then the electrode was placed into the cannula. Electrical stimulation at a frequency of 50 Hz was given for sensory testing after 300 to 700 ohms of impedance values were observed.

Paresthesia was questioned asking patients whether there is any pressure, compression or increase in pain where the needle tip was while testing. We accepted that the cannula is in the right place when paresthesia occurs below 0.5V. Motor stimulation was given with a frequency of 2 Hz. Motor response did not occur above 1.5 V. RF procedure was started after our location also confirmed by fluoroscopy. Pulse RF current at 42 °C at 20 ms 2 times per second was performed to patients for 360 seconds. The electrode was removed and needle entry site was closed with a sterile spunch after procedure completed. Patients were discharged within 6 hours .

Sample size calculation The sample size calculation was done using G*Power version 3.1.9.2 Software. Effect size f=0.25, α err prob=0.05, Power (1-β err prob)=0.80, Number of groups=2, Corr among rep measures=0.17, Noncentrality parameter λ=8.396, Critical F=4.007, Numerator df=1, Denominator df=58, Total sample size=60, Actual power= 0.813.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as having symptomatic lumbar disc prolapse based on the following:

  1. Clinical evidence of disc pulge in the form of disc related radicular pain of >3 months duration, not responding to conservative treatment and interfering with daily activities
  2. Radiological demonstration of posterolateral lumbar disc pulge by MRI lumbosacral
  3. Age range is between 30-80 years

Exclusion Criteria:

1. Patients with spinal deformities
2. Patients with a previous history of spinal trauma
3. Patients with previous spinal surgery
4. Patients with radiological evidence of any inflammatory or neoplastic lesion affecting the spinal cord or vertebral column
5. Patients with severe lumbar disc herniation causing lower limb weakness or sphincteric troubles
6. Patient with pain rather than radicular neuropathic pain as Facet osteoarthritis, Sacroiliitis, Hip osteoarthritis, Discogenic, Pyriformis syndrome.
7. Patients with contraindications to interventions (coagulopathy, sepsis, or allergy to the used drugs)
8. Patients with contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body).
9. Pregnant
10. History of G6PD deficiency in patients who are candidates to receive ozone therapy.
11. Suspected spondylodiscitis.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Modified Oswestry Back Disability Score | 3 months
  Functional disability
Numeric Rating Scale | 3 months
  Pain intensity
The Short Assessment of Patient Satisfaction | 3 months
  Patient's satisfaction

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mona Hussein, Banī Suwayf, Beni Suweif Governorate
  - Beni-Suef University, Banī Suwayf

IPD SHARING:
Plan to Share IPD: No